CLINICAL TRIAL: NCT01557166
Title: Effect of Liraglutide in Obese Subjects With Moderate or Severe Obstructive Sleep Apnoea. A 32 Week Randomised, Double-blind, Placebo-controlled, Parallel Group, Multi-centre and Multinational Trial
Brief Title: Effect of Liraglutide in Obese Subjects With Moderate or Severe Obstructive Sleep Apnoea: SCALE™ - Sleep Apnoea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-3970; U1111-1126-6260 (Other: WHO)
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Metabolism and Nutrition Disorder; Obesity; Obstructive Sleep Apnoea
Keywords: OSA
MeSH Terms: conditions — Nutrition Disorders; Obesity; Sleep Apnea, Obstructive | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide 3.0 mg (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — 3.0 mg liraglutide administered subcutaneously (s.c., under the skin) once daily for 32 weeks + diet and exercise
  Arms: Liraglutide 3.0 mg
Drug: placebo — Placebo administered subcutaneously (s.c., under the skin) once daily for 32 weeks + diet and exercise
  Arms: Placebo

SUMMARY:
This trial is conducted in North America. The aim of the trial is to investigate the effect of liraglutide in obese subjects with sleep apnoea.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Body mass index equal to or above 30 kg/m^2
* Stable body weight (less than 5% self-reported change during the previous 3 months)
* Diagnosis of moderate or severe obstructive sleep apnoea (OSA)
* Unwilling or unable to use continuous positive airway pressure (CPAP) (or other positive airway pressure) treatment. No CPAP (or other positive airway pressure) treatment for at least four weeks prior to screening
* Ability and willingness to comply with all protocol procedures e.g. correct handling of trial product, compliance to visit schedule and dietary advice and complete trial related questionnaires

Exclusion Criteria:

* Treatment with glucagon-like peptide-1 (GLP-1) receptor agonists, dipeptidyl peptidase-4 inhibitors or insulin within the last 3 months prior to screening
* Diagnosis of type 1 or type 2 diabetes per judgement of the investigator
* Glycosylated haemoglobin (HbA1c) equal to or above 6.5%
* Significant craniofacial abnormalities that may cause OSA
* Respiratory and neuromuscular diseases that could interfere with the results of the trial in the opinion of the investigator
* Use of central stimulants, hypnotics, mirtazepine, opioids, trazodone within the previous 3 months prior to screening
* Obesity induced by drug treatment
* Treatment with pramlintide, sibutramine, orlistat, zonisamide, topiramate or phenteremine within the last 3 month prior to screening
* Previous surgical treatment for obesity
* Screening calcitonin equal to or above 50 ng/L
* Familial or personal history of Multiple Endocrine Neoplasia type 2 or familial Medullary Thyroid Carcinoma
* Personal history of non-familial Medullary Thyroid Carcinoma
* History of chronic pancreatitis or idiopathic acute pancreatitis
* History of Major Depressive Disorder or suicide attempts
* Systolic blood pressure equal to or above 160 mmHg and/or diastolic blood pressure equal to or above 100 mmHg

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 359 (Actual)
Dates: Start 2012-06-07 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (36):
- United States (33):
  - Novo Nordisk Investigational Site, Glendale, California
  - Novo Nordisk Investigational Site, Oceanside, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Redwood City, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Santa Monica, California
  - Novo Nordisk Investigational Site, Brandon, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, South Miami, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Macon, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Vernon Hills, Illinois
  - Novo Nordisk Investigational Site, Overland Park, Kansas
  - Novo Nordisk Investigational Site, Crestview Hills, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Chevy Chase, Maryland
  - Novo Nordisk Investigational Site, North Dartmouth, Massachusetts
  - Novo Nordisk Investigational Site, Portage, Michigan
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Dublin, Ohio
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Warwick, Rhode Island
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Vienna, Virginia
- Canada (3):
  - Novo Nordisk Investigational Site, Burlington, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario

REFERENCES:
- [Result] O'Neil PM, Garvey WT, Gonzalez-Campoy JM, Mora P, Ortiz RV, Guerrero G, Claudius B, Pi-Sunyer X; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. EFFECTS OF LIRAGLUTIDE 3.0 MG ON WEIGHT AND RISK FACTORS IN HISPANIC VERSUS NON-HIPANIC POPULATIONS: SUBGROUP ANALYSIS FROM SCALE RANDOMIZED TRIALS. Endocr Pract. 2016 Nov;22(11):1277-1287. doi: 10.4158/EP151181.OR. Epub 2016 Aug 2. PMID 27482610
- [Result] Bays H, Pi-Sunyer X, Hemmingsson JU, Claudius B, Jensen CB, Van Gaal L. Liraglutide 3.0 mg for weight management: weight-loss dependent and independent effects. Curr Med Res Opin. 2017 Feb;33(2):225-229. doi: 10.1080/03007995.2016.1251892. Epub 2016 Nov 6. PMID 27817208
- [Result] Blackman A, Foster GD, Zammit G, Rosenberg R, Aronne L, Wadden T, Claudius B, Jensen CB, Mignot E. Effect of liraglutide 3.0 mg in individuals with obesity and moderate or severe obstructive sleep apnea: the SCALE Sleep Apnea randomized clinical trial. Int J Obes (Lond). 2016 Aug;40(8):1310-9. doi: 10.1038/ijo.2016.52. Epub 2016 Mar 23. PMID 27005405
- [Result] Steinberg WM, Rosenstock J, Wadden TA, Donsmark M, Jensen CB, DeVries JH. Impact of Liraglutide on Amylase, Lipase, and Acute Pancreatitis in Participants With Overweight/Obesity and Normoglycemia, Prediabetes, or Type 2 Diabetes: Secondary Analyses of Pooled Data From the SCALE Clinical Development Program. Diabetes Care. 2017 Jul;40(7):839-848. doi: 10.2337/dc16-2684. Epub 2017 May 4. PMID 28473337
- [Result] O'Neil PM, Aroda VR, Astrup A, Kushner R, Lau DCW, Wadden TA, Brett J, Cancino AP, Wilding JPH; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. Neuropsychiatric safety with liraglutide 3.0 mg for weight management: Results from randomized controlled phase 2 and 3a trials. Diabetes Obes Metab. 2017 Nov;19(11):1529-1536. doi: 10.1111/dom.12963. Epub 2017 Jul 21. PMID 28386912
- [Result] Davies MJ, Aronne LJ, Caterson ID, Thomsen AB, Jacobsen PB, Marso SP; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. Liraglutide and cardiovascular outcomes in adults with overweight or obesity: A post hoc analysis from SCALE randomized controlled trials. Diabetes Obes Metab. 2018 Mar;20(3):734-739. doi: 10.1111/dom.13125. Epub 2017 Nov 1. PMID 28950422
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 40 sites in 2 countries, as follows: United States: 35 sites; Canada: 5 sites.
Pre-assignment Details: The trial consisted of a 2-week screening period before randomisation.
Groups:
- Liraglutide 3.0 mg: Subjects were administered 3.0 mg of liraglutide subcutaneously (s.c., under the skin) once daily for 32 weeks. Subjects were also prescribed a 500 kcal/day-deficit diet and exercise for a minimum of 150 min/week.
- Placebo: Subjects were administered placebo subcutaneously (s.c., under the skin) once daily for 32 weeks. Subjects were also prescribed a 500 kcal/day-deficit diet and exercise for a minimum of 150 min/week.
Period: Overall Study
Arm/Group | Liraglutide 3.0 mg | Placebo
Started | 180 | 179
Exposed | 176 | 179
Completed | 134 | 142
Not Completed | 46 | 37
Not completed — Adverse Event | 20 | 6
Not completed — Lack of Efficacy | 2 | 1
Not completed — Protocol Violation | 8 | 5
Not completed — Withdrawn consent | 12 | 20
Not completed — Target dose not tolerated | 1 | 0
Not completed — Psychiatric disorder | 1 | 0
Not completed — Unclassified | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide 3.0 mg | Placebo | Total
Number analyzed (Participants) | 180 | 179 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (9.9) | 48.4 (9.5) | 48.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 50 | 101
  Male | 129 | 129 | 258
Body weight [Mean (Standard Deviation); unit: kg] | 116.5 (23.0) | 118.7 (25.4) | 117.6 (24.2)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 38.9 (6.4) | 39.4 (7.4) | 39.1 (6.9)
Apnoea-hypopnoea index (AHI) [Mean (Standard Deviation); unit: events/hour] | 49.0 (27.5) | 49.3 (27.5) | 49.2 (27.4)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 5.4 (0.6) | 5.4 (0.9) | 5.4 (0.8)
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] | 5.7 (0.4) | 5.6 (0.4) | 5.7 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Apnoea-hypopnoea Index (AHI)
Description: Observed mean change from baseline in AHI (events/hour) after 32 weeks of treatment. AHI (apnoea and hypopnoea events per hour of sleep) is a measure used for the diagnosis and severity classification of obstructive sleep apnoea. AHI severity category: none ≤4.9; mild 5.0-14.9; moderate 15.0-29.9; severe ≥30.0 events/hour.
Time Frame: Week 0, Week 32
Population: Full analysis set (FAS) - included all randomised subjects. 334 subjects contributed to the statistical analysis.
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 168 | 166
events/hour | -12.22 (23.34) | -6.08 (25.90)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; Let μ liraglutide 3.0mg and μ placebo denote mean change in AHI for liraglutide 3.0 mg and placebo,respectively. The null-hypothesis and the alternative was H0: μliraglutide 3.0mg = μplacebo against the alternative HA: μliraglutide 3.0mg ≠ μplacebo; Test type: Superiority or Other; p = 0.015, ANCOVA; ANCOVA model was used with treatment, country and sex as fixed factors, and the baseline value of AHI, baseline BMI and baseline age as covariates; Estimated treatment difference = -6.10, 95% CI [-11.0 to -1.19]

2. Secondary Outcome: Change From Baseline in Body Weight (kg)
Description: Observed mean change from baseline in fasting body weight (kg) after 32 weeks of treatment.
Time Frame: Week 0, week 32
Population: Full analysis set (FAS) - included all randomised subjects. 353 subjects contributed to the statistical analysis.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 175 | 178
kg | -6.73 (6.59) | -1.87 (5.44)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: Observed mean change from baseline in fasting plasma glucose (mmol/L) after 32 weeks of treatment.
Time Frame: Week 0, week 32
Population: Full analysis set (FAS) - included all randomised subjects. 355 subjects contributed to the statistical analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 178 | 177
mmol/L | -0.15 (0.69) | 0.17 (0.96)

4. Secondary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c) (%)
Description: Observed mean change from baseline in glycosylated haemoglobin (HbA1c) (%) after 32 weeks of treatment.
Time Frame: Week 0, week 32
Population: Full analysis set (FAS) - included all randomised subjects. 345 subjects contributed to the statistical analysis
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 174 | 171
percentage of glycosylated haemoglobin | -0.36 (0.30) | -0.17 (0.29)

ADVERSE EVENTS:
Time Frame: Events that either occur before randomisation and increase in severity during the treatment period or have an onset date on or after the first day of randomised treatment and no later than 14 days after the last day of randomised treatment.
Description: Safety analysis set - included all randomised subjects exposed to trial drug.
Arm/Group | Liraglutide 3.0 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 6/176 | 6/179
Other Adverse Events (participants affected / at risk) | 117/176 | 84/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 3.0 mg (N=176) | Placebo (N=179)
Angina pectoris (Cardiac disorders) | 2 (3) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1)
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 3.0 mg (N=176) | Placebo (N=179)
Constipation (Gastrointestinal disorders) | 21 (26) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 29 (38) | 14 (17)
Dyspepsia (Gastrointestinal disorders) | 15 (20) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (11) | 0 (0)
Nausea (Gastrointestinal disorders) | 47 (59) | 12 (14)
Vomiting (Gastrointestinal disorders) | 13 (16) | 5 (5)
Injection site haematoma (General disorders) | 7 (8) | 13 (14)
Influenza (Infections and infestations) | 9 (12) | 9 (9)
Nasopharyngitis (Infections and infestations) | 15 (19) | 18 (20)
Upper respiratory tract infection (Infections and infestations) | 18 (25) | 19 (25)
Lipase increased (Investigations) | 9 (11) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9)
Headache (Nervous system disorders) | 25 (26) | 20 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of plans by any investigator to publish and to review any scientific paper, presentation, communication or other information concerning the investigation described in the protocol. Novo Nordisk reserves the right to prior review of such publications and to ask for deferment of publication of individual site results until after the primary manuscript is accepted for publication.